CLINICAL TRIAL: NCT05834543
Title: Phase Ib Clinical Trial to Evaluate the Safety and Efficacy of TQB2618 Injection Combined Therapy in Patients With Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Clinical Trial to Evaluate the Safety and Effectiveness of TQB2618 Injection Combined Therapy in Patients With Advanced Esophageal Squamous Cell Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This study was closed due to business reasons. Closure was not prompted by any safety or efficacy concerns.
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB2618-AK105-Ib-03
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2024-10

CONDITIONS: Advanced Esophageal Squamous Cell Carcinoma
MeSH Terms: interventions — penpulimab; Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TQB2618 injection +Penpulimab injection+Chemotherapy (Experimental): Experimental group in Cohort 1. TQB2618 injection, Penpulimab injection, Paclitaxel, Cisplatin, 21 days as a treatment cycle. After 4~6 cycles, TQB2618 injection combined Penpulimab injection, 21 days as a treatment cycle.
  Interventions: Drug: TQB2618 injection, Penpulimab injection, Paclitaxel, Cisplatin
- Penpulimab injection+Chemotherapy (Active Comparator): Active comparator group in Cohort 1. Penpulimab injection, Paclitaxel, Cisplatin, 21 days as a treatment cycle.
  After 4~6 cycles, Penpulimab injection 21 days as a treatment cycle.
  Interventions: Drug: Penpulimab injection, Paclitaxel, Cisplatin
- TQB2618 injection +Penpulimab +TQB3617capsules (Experimental): Cohort 2. TQB2618 injection, Penpulimab injection, 21 days as a treatment cycle.
  TQB3617 capsules are administered on Day 1 and Day 14, 21 days as a treatment cycle.
  Interventions: Drug: TQB2618 injection, Penpulimab injection, TQB3617capsules

INTERVENTIONS:
Drug: TQB2618 injection, Penpulimab injection, Paclitaxel, Cisplatin — TQB2618 injection：Anti-TIM-3 monoclonal antibody. Penpulimab injection：Humanized Monoclonal Antibody to Programmed Cell Death Protein 1 (PD-1).
  Paclitaxel and Cisplatin are chemotherapy.
  Arms: TQB2618 injection +Penpulimab injection+Chemotherapy
Drug: Penpulimab injection, Paclitaxel, Cisplatin — Penpulimab injection：Humanized Monoclonal Antibody to Programmed Cell Death Protein 1 (PD-1).
  Paclitaxel and Cisplatin are chemotherapy.
  Arms: Penpulimab injection+Chemotherapy
Drug: TQB2618 injection, Penpulimab injection, TQB3617capsules — TQB2618 injection：Anti-TIM-3 monoclonal antibody. Penpulimab injection：Humanized Monoclonal Antibody to Programmed Cell Death Protein 1 (PD-1).
  Arms: TQB2618 injection +Penpulimab +TQB3617capsules

SUMMARY:
To investigate the efficacy and safety of TQB2618 injection combined Penpulimab and chemotherapy in the first-line treatment of recurrent/metastatic esophageal squamous cell carcinoma compared with Penpulimab combined chemotherapy.

The primary efficacy outcomes are progression free survival (PFS) and objective response rate (ORR).

ELIGIBILITY:
Inclusion Criteria:

* Nonresectable locally advanced, recurrent or metastatic esophageal squamous cell carcinoma (excluding mixed adenosquamous cell carcinoma) confirmed by histopathology or cytology;
* For Cohort 1: Those who have not received systematic treatment, or have relapse at least 6 months after the (new) adjuvant treatment/radical radiotherapy and chemotherapy; For Cohort 2: received platinum-based chemotherapy and immuno checkpoint inhibitor (PD-1/PD-L1, etc.) treatment and failed, the best effect of front-line immunotherapy CR, PR, or SD lasted ≥ 24 weeks, and there was evidence of imaging progression;
* Age: 18-75 years old (calculated based on the date of signing the informed consent); Eastern Cooperative Oncology Group (ECOG) score: 0-1; The expected survival period is more than 3 months;
* At least one measurable lesion was confirmed according to RECIST 1.1 standard; Measurable lesions should not have received local treatment such as radiotherapy (lesions located in the area of previous radiotherapy treated can also be selected as target lesions if progression is confirmed);
* The main organs function well and meet the following standards:

  1. The blood routine examination should meet the following requirements: (no blood transfusion, no use of hematopoietic stimulator drugs for correction within 14 days before the examination)

     1. Hemoglobin content (HB) ≥ 90g/L;
     2. Absolute neutrophil count (ANC) ≥ 1.5 ×10^9/L；
     3. Platelet count (PLT) ≥ 100 × 10^9/L.
  2. Biochemical examination shall meet the following standards:

     1. Total serum bilirubin (TBIL) ≤ 1.5 times of the upper limit of normal value (ULN);
     2. Alanine transaminase (ALT) and aspartate aminotransferase (AST) ≤ 2.5ULN; In case of liver metastasis, ALT and AST ≤ 5ULN;
     3. Serum creatinine (Cr) ≤ 1.5ULN or creatinine clearance rate (CCr) ≥ 60ml/min; (Cockcroft-Default formula);
  3. Coagulation function is sufficient, defined as international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN;
  4. Thyroid function examination shall meet the following standards: thyroid stimulating hormone (TSH) ≤ ULN; If abnormal, exam the level of T3 and T4, patients with abnormal T3 and T4 can be enrolled.
  5. Cardiac color doppler evaluation: left ventricular ejection fraction (LVEF) ≥ 50%.
  6. Female subjects of childbearing age should agree to use contraceptives (such as intrauterine devices, contraceptives or condoms) during the study period and within 6 months after the end of the study; The serum pregnancy test was negative within 7 days before enrollment and must be a non-lactating subject; Male subjects should agree to use contraception during the study period and within 6 months after the end of the study.
  7. Subjects volunteered to join the study and signed the informed consent form, with good compliance;

Exclusion Criteria:

* Known esophageal squamous cell carcinoma which tended to complete obstruction under endoscope and needed interventional treatment to relieve obstruction;
* Increased risk of bleeding or fistula caused by tumor significantly invading adjacent organs (aorta or trachea);
* After esophageal or tracheal stent implantation;
* For Cohort 1: Patients who have used paclitaxel in adjuvant chemotherapy and have relapse or metastasis within one year (note: those who have relapse or metastasis for more than one year can be included in the study); Patients who received cisplatin dose ≥ 300mg/m2 in the year before;
* The load of liver metastases accounts for more than 50% of the whole liver volume;
* For Cohort 1: Those who have received anti-PD-1 or anti-PD-L1/PD-L2, TIM-3, CTLA-4 drugs or other therapies that act on T-cell co-stimulation targets or checkpoints in the past; For Cohort 2: Patients who have previously received BET inhibitor treatment.
* Patients with any serious and/or uncontrollable diseases, including:

  1. Have any clinical cardiovascular symptoms or diseases with poor control, including but not limited to: patients with poor blood pressure control using antihypertensive drugs (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg); New York Heart Association (NYHA) grade II or above heart failure; Unstable angina pectoris; Myocardial infarction occurred in the past one year; Patients with arrhythmia (QTc ≥ 450ms (male), QTc ≥ 470ms (female)), or patients with left ventricular ejection fraction (LVEF)<50% according to cardiac color Doppler examination;
  2. Active or uncontrolled serious infection (≥ NCI CTC AE level 2 infection);
  3. Liver diseases such as cirrhosis, decompensated liver disease, chronic active hepatitis (hepatitis B virus (HBV) reference: HBsAg positive, and HBV DNA detected value exceeds the upper limit of normal value; hepatitis C virus (HCV) reference: HCV antibody positive, and HCV virus titer detected value exceeds the upper limit of normal value); Note: Subjects with positive hepatitis B surface antigen or core antibody and hepatitis C patients who meet the inclusion conditions need to receive continuous antiviral treatment to prevent virus activation.
  4. Poor control of diabetes (Fasting Blood Glucose (FBG)>10mmol/L);
  5. Urine routine test showed that urine protein ≥++, and confirmed that the 24-hour urine protein content was more than 1.0 g;
  6. Renal failure requiring hemodialysis or peritoneal dialysis;
  7. Those who have epilepsy and need treatment;
* Major surgery (craniotomy, thoracotomy or laparotomy) has been performed within 4 weeks before the first dose of the study or is expected to require major surgery during the study treatment.
* A history of gastrointestinal perforation and/or fistula within 6 months before treatment; Or have experienced arterial/venous thrombosis events, such as cerebrovascular accident (including transient ischemic attack), deep venous thrombosis and pulmonary embolism;
* Known central nervous system metastasis and/or cancerous meningitis;
* Ascites with clinical significance, including any ascites that can be found in physical examination. For ascites that have been treated in the past or still need to be treated at present, subjected can be included if only a small amount of ascites is shown by imaging and without symptoms;
* Patients with equal amount of effusion in both sides of the chest, or a large amount of effusion in one side of the chest, or who have caused respiratory dysfunction and need drainage;
* Wounds or fractures that have not been cured for a long time;
* Esophageal squamous cell carcinoma patients with active bleeding of the primary lesion within 2 months; Pulmonary hemorrhage with NCI CTC AE grade>1 occurred within 4 weeks before enrollment; Bleeding at other sites with NCI CTC AE grade>2 occurred within 4 weeks before enrollment; Patients with bleeding tendency (such as active gastrointestinal ulcer) or undergoing thrombolytic or anticoagulant therapy such as warfarin, heparin or its analogues;
* There is active pulmonary tuberculosis, or there is a history of active tuberculosis infection within one year before enrollment, or there is a history of active tuberculosis infection more than one year before enrollment, but they have not received treatment;
* Interstitial lung disease requiring steroid hormone treatment;
* Uncontrolled metabolic disorder or other non-malignant tumor organ or systemic disease or cancer secondary reaction, which may lead to higher medical risk and/or uncertainty of survival evaluation;
* Patients with significant malnutrition (such as the need for continuous parenteral nutrition ≥ 7 days), patients with Body Mass Index（BMI）<18.5kg/m2 or weight loss ≥ 10% in the two months before screening.
* Those who have a history of abuse of psychotropic substances and are unable to quit or have mental disorders;
* Have a history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation and hematopoietic stem cell transplantation;
* History of other primary malignant tumors, except for the following: 1) Malignant tumors completely relieved for at least 2 years before enrollment and no other treatment is required during the study period; 2) Nonmelanoma skin cancer or malignant freckle-like nevus with sufficient treatment and no evidence of disease recurrence; 3) Carcinoma in situ with sufficient treatment and no evidence of disease recurrence;
* Those who are allergic to the study drug or its excipients, or to similar drugs;
* Pregnant or lactating female patients;
* There is an unrelieved toxic reaction higher than NCI CTC AE level 1 caused by any previous treatment before the first medication, excluding hair loss;
* Active autoimmune diseases requiring systemic treatment (such as the use of disease relief drugs, corticosteroids or immunosuppressants) have occurred within 2 years before the first medication. Replacement therapy (such as thyroxine, insulin or physiological corticosteroids for adrenal or pituitary insufficiency) is not considered as systemic treatment;
* Have received systemic glucocorticoid therapy (dose>10mg/day prednisone or other effective hormones) or any other form of immunosuppressive therapy within 2 weeks before the start of the study;
* The history of live attenuated vaccine inoculation within 28 days before the first administration or the planned live attenuated vaccine inoculation during the study period;
* Have received chemotherapy, radiotherapy or other anti-tumor treatment within 4 weeks before the first medication (washout period is calculated from the end of the last treatment); Note: Those who have received local radiotherapy in the past can be enrolled if the following conditions are met: the end of radiotherapy is more than 3 weeks from the beginning of study treatment (brain radiotherapy is more than 2 weeks); And the target focus selected in this study is not in the radiotherapy area; Or the target lesion is located in the radiotherapy area, but progress has been confirmed.
* Participated in clinical trials of other anti-tumor drugs within 4 weeks before the first medication (the washout period is calculated from the end of the last treatment);
* Within 2 weeks before the first use of drug, the subjects have received the treatment of traditional Chinese medicines (including compound cantharides capsule, Kangai injection, Kanglaite capsule/injection, Aidi injection, Brucea javanica oil injection/capsule, Xiaoaiping tablet/injection, cinobufagin capsule, etc.) with anti-tumor indications specified in the drug labelling approved by National Medical Products Administration (NMPA).
* Subjects who, according to the judgment of the investigator, have serious concomitant diseases that endanger the safety of the patient or affect the completion of the study, or who are considered that are not suitable for enrollment due to other reasons .

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-05-26 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
PFS | Baseline up to two years.
  The time from the first administration of the drug to disease progression or death (whichever occurs first).
ORR | Baseline up to two years.
  According to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and iRECIST, the proportion of subjects whose tumors are evaluated as complete response(CR) and partial response(PR) by subcenter imaging evaluation. It is recorded from the first use of the drug to disease progression or initiation of a new anticancer treatment.

SECONDARY OUTCOMES:
Overall survival (OS) | Baseline up to death event, assessed up to 2 years.
  From randomization to the time of death from any cause.
Disease Control Rate (DCR) | Baseline to up to two years.
  The percentage of participants with complete response (CR), partial response (PR), or stable disease (SD) at 6 weeks or greater than or equal to as determined by investigators according to Response evaluation criteria in solid tumors (RECIST) 1.1.
Duration of Remission (DOR) | Baseline to up to two years.
  The period from firstly-recorded objective tumor response (CR or PR) to firstly-recorded objective tumor progression or death due to any cause (whichever occurs first).
Incidence of adverse events (AEs) | Baseline to up to two years.
  All adverse medical events that occur after the subject receives the investigational drug may be manifested as symptoms, signs, disease, or laboratory abnormalities, but are not necessarily causally related to the investigational drug. The adverse events were evaluated according to the National Cancer Institute standard for common toxic reactions (NCI-CTC v5.0).
Severity of adverse events (AEs) | Baseline to up to two years.
  All adverse medical events that occur after the subject receives the investigational drug may be manifested as symptoms, signs, disease, or laboratory abnormalities, but are not necessarily causally related to the investigational drug. The severity of adverse events were evaluated according to the National Cancer Institute standard for common toxic reactions (NCI CTC) V5.0.
Incidence of serious adverse events (SAEs) | Baseline to up to two years.
  It refers to adverse medical events such as death, life-threatening, permanent or serious disability or loss of function, hospitalization or prolonged hospitalization, and congenital abnormalities or birth defects after the subject receives the experimental drug.

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Tongling People's Hospital, Tongling, Anhui
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - AnYang Tumor Hospital, Anyang, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Zhumadian Central Hospital, Zhumadian, Henan
  - Affiliated Hospital of Jining Medical College, Jining, Shandong
  - Changzhi People's Hospital, Changzhi, Shanxi
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi, Shanxi
  - Jincheng General Hospital, Jincheng, Shanxi